CLINICAL TRIAL: NCT07130071
Title: A Pragmatic, Stepped Wedge, Multi-centre, Cluster Randomised Trial Evaluating the Efficiency of Algorithm Technology and Tailored Primary Care Quality Improvement Support to Identify, Diagnose and Refer Patients With Rare and Difficult to Diagnose Disease (Defined by the NHS as Those Suffering From Significant Diagnostic Odyssey)
Brief Title: Channelling Algorithm Proficiency To Understand, Recognise and Elucidate Disease
Acronym: CAPTURED
Status: Not yet recruiting | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Responsible Party: Sponsor
Other Study IDs: OPRIUK-2102
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Rare Disorders
Keywords: rare disease; rare disorder; difficult to diagnose; quality improvement; algorithm
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GP practices with patients identified by one of the QIP algorithms.: GP practices are the participants of the trial and not individual patients. We will invite GP practices to take part in the trial. Algorithms will be run on an anonymised dataset, OPCRD, to identify practices with high-risk patients. Practices that wish to participate and meet the trial eligibility criteria will be required to sign Clinical Trial Agreements.

SUMMARY:
Rare diseases affect over 3.5 million people in the UK. It can take years of multiple referrals, inconclusive tests or incorrect diagnoses, for patients to get a final diagnosis. We call this diagnostic odyssey, and GPs are often the first point of call for patients at the start.

Algorithms can be used to help identify patients with rare diseases faster, who may benefit from testing. They also help healthcare professionals in decision making. Healthcare providers also recognise the value of quality improvement (QI) activities, but practices are often reluctant to participate in non-QOF QI initiatives.

CAPTURED aims to help reduce the diagnostic odyssey patients face by evaluating the efficiency of algorithms and tailored primary care QI support to identify, diagnose and refer patients with rare and difficult to diagnose disease. It will contribute towards these aspects of the UK Rare Disease Framework: (Priority 1) helping patients get a final diagnosis faster; and (Priority 2) increasing awareness of rare diseases among healthcare professionals.

CAPTURED will run as a stepped wedge, cluster randomised trial. Practices are the participants, and not individual patients. Practices will be randomly allocated to undertake quality improvement programmes (QIP) to help evaluate up to 10 rare disease algorithms. Practices will undertake QIPs at specific times, but at the end, all practices would undertake all the QIPs they have at-risk patients for. Practices will invite at-risk patients for testing/screening, and refer newly diagnosed patients for appropriate care. Practices will be supported with the QIPs by OPC Quality Improvement and Research Support Service, at no cost to practices.

CAPTURED will run for 5 years and will enrol 500 practices. The trial does not involve any medicine, drug or equipment. The trial will use anonymised patient data collected from all participating practices into the Optimum Patient Care Research Database (OPCRD).

DETAILED DESCRIPTION:
The aim of CAPTURED is to evaluate the efficiency of algorithm technology and tailored primary care quality improvement support in identifying, testing and referring patients at high probability of specific rare or difficult to diagnose disease.

The trial aims to reduce the diagnostic odyssey for rare and difficult to diagnose disease patients and facilitate quicker access to appropriate treatment, utilising algorithms designed to identify patients that are at high probability.

CAPTURED is a series of quality improvement programs (QIPs) that are each delivered in a stepped wedge model, to enable comparison between the QI intervention and standard care. Each QIP, under CAPTURED, will utilise a specific algorithm for rare or difficult to diagnose disease, and a specific diagnostic testing/quality improvement support package. It is planned to run for 5 years (2025-2030). Each QIP will run for a defined period.

CAPTURED is UK-wide multicentre study. All participating practices should be able to accept the intervention (diagnostic test/screening and tailored quality improvement support package) as part of their patient care. CAPTURED will be conducted at an estimated 500 GP practices in the UK. Only practices with patients identified as at high probability of specific rare or difficult to diagnose disease will participate in each project. The algorithms use digital biomarkers in patients electronic medical record data such as symptoms, diagnoses and healthcare utilisation to identify patients who would benefit from specific diagnostic testing. Individual projects will have specific cut-offs to determine high probability of disease but typically it is a likelihood of 60% or more.

Practices with patients with high probability of disease will be randomised into clusters. Randomisation will occur individually for each QIP. The intervention (diagnostic testing/screening and quality improvement support package) will be given at different time-points defined by the stepped wedge design.

The index date (time = 0) will be defined as the date that the first cluster of practices receives communication about having patients identified as at high probability of rare or difficult to diagnose disease. Communication with remaining clusters will be sent out at the exact time points defined by the stepped wedge design but will be specific to each project.

The primary objective of CAPTURED is to demonstrate that the patient testing pathway works defined as:

• To determine if algorithm technology and quality improvement support increases rates of diagnosis of rare or difficult to diagnose disease.

The secondary objectives of the trial are outlined below:

* To determine if the algorithm technology and quality improvement support improves rates of diagnostic testing for patients at high probability of rare or difficult to diagnose disease.
* To evaluate the efficacy of communication with patients regarding the quality improvement intervention.
* To evaluate the rate of acceptance of the quality improvement intervention in the eligible patient population.

The following exploratory objectives will be explored as part of the trial:

* To evaluate if the algorithms identify suitable patients as high probability for rare or difficult to diagnose disease, who are deemed clinically appropriate for further testing by Medical professional judgement .
* To evaluate the outcomes of the diagnostic testing with regard to alternative diagnosis being derived as a direct result of the quality improvement programmes.

Results for all projects (up to 10) will be combined for overall analysis of CAPTURED at the end of the 5-year planned trial period.

The algorithm for each QIP will be run at baseline on the Optimum Patient Care Research Database (OPCRD) and the Optimum Patient Care Research Database (OPCSD), to identify practices with patients who are at high probability of disease. Only practices (and their patients) that fulfil the inclusion criteria and none of the exclusion criteria will be included. Initially, practices with a population of at least 15,000 patients will be included, to maximise likelihood of identifying patients at high probability of disease. This is a flexible cut-off that can be removed depending on numbers of patients identified. Practices that have no current high probability patients for a particular QIP will be excluded from that QIP only but will remain in the CAPTURED overarching trial and eligible for further QIPs.

Participating practices will be offered quality improvement support which will include specific diagnostic testing. Exact details of quality improvement support provided will be determined by each QIP and will all comprise the following core activities:

1. Identification (using algorithm)
2. Medical review of patients (EHR data) and/or expert review of patients
3. Provision of test/screen to patients
4. Guidance and support/assistance with patient referrals and follow-on care

These are patient care activities and are NOT research activities.

The specific diagnostic testing process may be remote (e.g. delivered to patients), at practice or at a specified test centre; and will be determined by each QIP.

Once testing has been completed, the patient and GP practice are informed of the result and supported with further steps, as required. Anonymised patient data from participating practices will be collected for trial analysis.

Evaluation of CAPTURED will occur at the end of the 5-year study period.

Practices will be considered as in the control phase in the pre-intervention window. Once randomisation occurs practices move from control to intervention at different points in time. So, all practices contribute some data to both control and intervention periods. Thus, the comparison is those control periods versus those intervention periods.

The proposed study population will be GP practices with patients flagged by the algorithm(s) in the Optimum Patient Care Research Database (OPCRD) and the Optimum Patient Care Service Database (OPCSD). The OPCRD is a REC approved, longitudinal electronic medical record database of over 29 million patients in the UK that is established and managed by Optimum Patient Care Ltd (OPC). OPCSD is pseudonymised patient database used to provide ongoing quality improvement services and programmes to GP practices across the UK.

ELIGIBILITY:
Inclusion Criteria:

* General practice in the United Kingdom (England, Scotland, Wales, Northern Ireland) participating in Optimum Patient Care services and contributing deidentified data to OPCRD.
* At least 1 patient identified as high probability of rare or difficult to diagnose disease by one of the quality improvement program algorithms.

Exclusion Criteria:

* General practices hosting or affected by research, or other aspects of care, which might significantly influence the implementation of CAPTURED.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 500 practices will be recruited into the CAPTURED trial. The proposed study population will be GP practices with patients identified by the algorithm(s) in the Optimum Patient Care Research Database (OPCRD) and the Optimum Patient Care Service Database (OPCSD). The OPCRD is a REC approved, longitudinal electronic medical record database of over 29 million patients in the UK that is established and managed by Optimum Patient Care Ltd (OPC). OPCSD is pseudonymised patient database used to provide ongoing quality improvement services and programmes to GP practices across the UK.
  A total of 500 practices will be recruited into the CAPTURED trial.
  CAPTURED will be delivered in collaboration with Optimum Patient Care Ltd (OPC), as part of quality improvement and research support services provided to each participating GP practices with data collection into OPCSD (for QI and patient care) and OPCRD(for ethically approved research).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients given diagnosis for rare or difficult to diagnose disease | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Rate of patients given diagnosis for rare or difficult to diagnose disease in intervention population compared to rate of patients given diagnosis for rare or difficult to diagnose disease in control population, in a comparable time frame who receive delayed roll out, by way of a step wedge implementation .
  Definition: Direct comparison between (1) Total number of patients who are positively diagnosed as a direct result of the intervention in the intervention population/whole patient population for intervention population and (2) Total number of patients who are positively diagnosed in the control population/whole patient population for the control population.

SECONDARY OUTCOMES:
Rate of patients successfully completing diagnostic testing/screening | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Rate of patients successfully completing diagnostic testing/screening in intervention population compared to control population, in a comparable time frame who receive delayed roll out, by way of a step wedge implementation .
  Definition: Direct comparison between (1) Total number of patients who successfully complete diagnostic testing as a direct result of the intervention in the intervention population and (2) Total number of patients who successfully complete diagnostic testing in control population in a comparable time frame who receive delayed roll out, by way of a step wedge implementation .
Rate that patients are successfully contacted about testing/screening. | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Rate that patients are successfully contacted about testing/screening = total number of patients identified by the algorithm who are successfully contacted about testing/screening / number of patients identified by the algorithm deemed eligible for testing after practice and medical review.
Rate that patients are agreeing to testing/screening for rare or difficult to diagnose disease. | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Rate that patients agree to testing/screening = total number of patients identified by the algorithm who are successfully contacted about testing/screening AND agree to testing or screening/number of patients identified by the algorithm with who attempted contact is made.

OTHER OUTCOMES:
Proportion of patients the algorithm identified as high probability of rare or difficult to diagnose disease deemed clinically appropriate for testing, defined by Medical professional judgement. | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Proportion of patients the algorithm identified deemed clinically appropriate for testing, defined by Medical professional judgement = number of patients identified by algorithm as high-risk deemed clinically appropriate for testing following review by Medical Professional/number of patients identified by the algorithm as high-risk that undergo review by Medical professional.
Results of testing (regardless of outcome-positive, negative and alternative diagnosis). | Each individual QIP will have a defined time-frame as per the stepped-wedge design. Anonymised data of patients will be collected throughout the project for each participating practice. Results will be analysed at the end of the 5-year trial period.
  Results of diagnostic testing will be recorded, regardless of result. This will include positive and negative results for specific diseases that the algorithm is identifying patients for and also any alternative diagnoses derived from the quality improvement process.

CONTACTS AND LOCATIONS:
Overall Officials: Ursie Smith, PhD MBChB MSci Bsc, Principal Investigator — Observational and Pragmatic Research Institute (OPRI); David Price, MD PhD, Principal Investigator — Observational and Pragmatic Research Institute (OPRI)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for CAPTURED trial — https://www.opri.org.uk/captured
- See also: Website for Optimum Patient Care Research Database — https://opcrd.optimumpatientcare.org/
- See also: Website for Observational and Pragmatic Research Institute — https://www.opri.org.uk/